CLINICAL TRIAL: NCT06178523
Title: Cost-effective Treatment of Unexplained Infertility: A Prospective Multicenter, Double-blinded, Randomised Controlled Study
Brief Title: Cost-effective Treatment of Unexplained Infertility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Batterjee Medical College (Other)
Responsible Party: Principal Investigator, Remah Moustafa Kamel, Professor of Obstetrics and Gynaecology, Batterjee Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RES/2024/1
Record Dates: First submitted 2023-08-27; First posted 2023-12-21 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Unexplained Infertility
Keywords: Clomiphene citrate; Sildenafil citrate; Intrauterine insemination; Unexplained Infertility
MeSH Terms: interventions — Clomiphene; Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: Couples with unexplained infertility (n=900) were divided into three equal groups. Group-A received Sildenafil Citrate (Viagra®) and Clomiphene Citrate (Clomid®). Group-B received Clomiphene Citrate (Clomid®) and subjected to intra-uterine insemination (IUI). Group-C received Clomiphen Citrate (Clomid®) alone (Control group).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double (Clinical investigator; the Radiologist, and Biostatistician; data analyst).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Sildenafil & Clomiphene Group (Active Comparator): Sildenafil Acetate (Viagra®) 25 mg as a vaginal tablet 6 hourly for 10 days starting from the fifth day of the menstrual cycle + Clomiphene Citrate (Clomid®) 100 mg for 5 days starting from the second day of the menstrual cycle.
  Follow-up by resistance index (RI), pulsatility index (PI), and maximum velocity (T-max) of sub-endometrial, uterine, and ovarian vessels measured by using TVS Colour Doppler ultrasound.
  Interventions: Drug: Clomiphene Citrate.; Drug: Sildenafil Citrate
- IUI & Clomiphene Group (Active Comparator): Clomiphene Citrate (Clomid®) 100 mg for 5 days starting from the second day of the menstrual cycle + Intrauterine insemination (IUI) 42 hours after human chorionic gonadotropin (Pregnyl®) 10,000 IU injection IM.
  Follow-up by resistance index (RI), pulsatility index (PI), and maximum velocity (T-max) of sub-endometrial, uterine, and ovarian vessels measured by using TVS Colour Doppler ultrasound.
  Interventions: Drug: Clomiphene Citrate.; Procedure: Intrauterine Insemination
- Clomiphene only Group (Placebo Comparator): Clomiphene Citrate (Clomid®) 100 mg for 5 days starting from the second day of the menstrual cycle.
  Follow-up by resistance index (RI), pulsatility index (PI), and maximum velocity (T-max) of sub-endometrial, uterine, and ovarian vessels measured by using TVS Colour Doppler ultrasound.
  Interventions: Drug: Clomiphene Citrate.

INTERVENTIONS:
Drug: Clomiphene Citrate. — Clomiphene Citrate (Clomid®) 100 mg for 5 days starting from the second day of the menstrual cycle (Groups A, B, and C).
  Other Names: Clomid®
Drug: Sildenafil Citrate — Sildenafil Acetate (Viagra®) 25 mg as a vaginal tablet 6 hourly for 10 days starting from the fifth day of the menstrual cycle (Group-A).
  Other Names: Viagra®
  Arms: Sildenafil & Clomiphene Group
Procedure: Intrauterine Insemination — IUI (Group-B).
  Other Names: IUI
  Arms: IUI & Clomiphene Group

SUMMARY:
The issue of unexplained infertility that Southam brought up in 1960 is still a problem today. Despite improvements in infertility assessment, many couples still don't know why they are infertile. Even with the use of the most advanced ovulation detectors, fallopian tube patency tests, and semen evaluations, competency cannot identify every potential flaw in the intricate processes leading to conception. Unexplained infertility will be a challenge for both biological and clinical researchers since it results from these gaps in our understanding of fertilization and from our incapacity to use all of the current evidence-based information.

DETAILED DESCRIPTION:
For the treatment of unexplained infertility, Clomiphene Citrate (CC) is frequently used either alone or in conjunction with intrauterine insemination (IUI). Its combined oestrogenic and anti-oestrogenic characteristics serve as the basis for the mechanism of action. When clomiphene citrate is used, the uterine blood flow is reduced during the peri-implantation stage of early luteal phase. About 80% of women experience ovulation, which has a cumulative effect over 6 to 8 months, yet the pregnancy rate in these women can still be relatively low. The endometrial and cervical mucus-level anti-oestrogenic actions of CC are the potential culprits. Without a doubt, one of the biggest obstacles in treating infertility is the endometrial impact. If the endometrial thickness (ET) is less than 6 mm, the pregnancy rate may be extremely low.

Sildenafil citrate promotes endometrial thickness and uterine blood flow. The capacity of the blastocyst to penetrate the endometrium and establish a lasting blood supply is crucial for successful implantation. To do this, the blastocyst needs genes in order to create the required proteins for breaking down the endometrial cellular matrix, control cell development, and trigger angiogenesis.

It can be difficult to understand the evidence on the efficacy and security of therapy for unexplained infertility. Given the substantial proportion of unaided pregnancies with expectant management, it is problematic that most studies do not include a placebo or untreated control group.

ELIGIBILITY:
Inclusion Criteria:

* Saudi women.
* Married women in a stable, continuous, unprotected heterosexual relationship (cohabitating with their husbands).
* Aged between 18 to 35 years old.
* Non-smoking.
* Non-alcohol drinking.
* With a body mass index < 30 Kg/M2,
* Who are looking healthy (all their infertility-workup investigations including male partners' seminal analysis were within normal range)
* Failed to conceive spontaneously within 2 years of marriage without evident cause (cases with primary infertility).

Exclusion Criteria:

* All non-Saudi women,
* Saudi unmarried women (not yet engaged in sexual activity),
* Married women with age less than 18 or more than 35 years old,
* Patients with secondary infertility,
* Cigarette smokers.
* Alcohol drinking.
* BMI > 30 Kg/M2,
* Pregnant women.
* Breastfeeding women.
* With known pathological cause (either male or female factor),
* With hypersensitivity to any of medication planned to be used in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females with unexplained infertility.
Enrollment: 900 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcome | 7 weeks after positive pregnancy test.
  Ultrasound confirmation of intrauterine fetal heartbeat.

CONTACTS AND LOCATIONS:
Overall Officials: Remah M Kamel, PhD, Principal Investigator — Batterjee Medical College
Locations (1):
- Batterjee Medical College, Jeddah, Mecca Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No